CLINICAL TRIAL: NCT03704441
Title: ED50 and ED95 of Intrathecal Hyperbaric Bupivacaine With Fentanyl for Transurethral Prostatectomy in Elderly Patients : a Prospective Double-blinded Randomized Trial
Brief Title: ED50 and ED95 of Intrathecal Hyperbaric Bupivacaine With Fentanyl for Transurethral Prostatectomy in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KangnamAnes
Record Dates: First submitted 2018-08-01; First posted 2018-10-12 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2020-04

CONDITIONS: Old Age
Keywords: Spinal anesthesia in old age
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- bupivacaine 6mg (Other): bupivacaine 6mg
  Interventions: Drug: Bupivacaine
- bupivacaine 7mg (Other): bupivacaine 7mg
  Interventions: Drug: Bupivacaine
- bupivacaine 8mg (Other): bupivacaine 8mg
  Interventions: Drug: Bupivacaine
- bupivacaine 9mg (Other): bupivacaine 9mg
  Interventions: Drug: Bupivacaine
- bupivacaine 10mg (Other): bupivacaine 10mg
  Interventions: Drug: Bupivacaine
- bupivacaine 11mg (Other): bupivacaine 11mg
  Interventions: Drug: Bupivacaine
- bupivacaine 12mg (Other): bupivacaine 12mg
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — bupivacaine dose

SUMMARY:
As people age, the incidence of prostate hyperplasia increases. So patients under Transurethral Resection of Prostate(TURP) or Holmium Laser Ennucleation of Prostate(HoLEP) are mostly ole age people. Most old age patient has several underlying disease. So patients can develop high mortality and morbidity. Most surgeries for Prostate Resection are taken under Spinal anesthesia. Adequate block level for Prostate Resection is T10. But sometimes, old age patients can develop severe complication after spinal anesthesia. So we started this study to know the adequate drug concentration for Spinal anesthesia taken for Prostate Resection surgery.

DETAILED DESCRIPTION:
As people age, the incidence of prostate hyperplasia increases. So patients under Transurethral Resection of Prostate(TURP) or Holmium Laser Ennucleation of Prostate(HoLEP) are mostly ole age people. Most old age patient has several underlying disease. So patients can develop high mortality and morbidity. Most surgeries for Prostate Resection are taken under Spinal anesthesia. Adequate block level for Prostate Resection is T10. But sometimes, old age patients can develop severe hypotension and vital unstability due to unintentional high sensory and motor blocks. These complications are due to the decreased cerebrospinal fluid volume with increase of age. So we started this study to know the adequate drug concentration for Spinal anesthesia taken for Prostate Resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for TURP & HoLEP under spinal anesthesia
* Male between 65 and 100
* The American Society of Anesthesiologists physical status class 1 or 2

Exclusion Criteria:

* Patients with coagulopathy
* Patients with infectious disease
* Patients with a drug allergy
* Patients under 50kg or over 100kg
* In case of switching to general anesthesia

Ages: 65 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
ED50 and ED95 of intrathecal hyperbaric bupivacaine with fentanyl for transurethral prostatectomy in elderly patients | 2years
  ED50(50% Effective dose) and ED95(95% Effective dose) of intrathecal hyperbaric bupivacaine with fentanyl for transurethral prostatectomy in elderly patients

SECONDARY OUTCOMES:
comparison of incidence of complications(hypotension, nausea/vomiting and shivering) during perioperative period | 2years
  comparison of incidence of complications(hypotension, nausea/vomiting and shivering) during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Eun Mi Choi, MD, Study Director — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam sacred heart hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No